CLINICAL TRIAL: NCT06646094
Title: Assessment of Cognitive Functions in Patients Receiving Whole Brain Radiotherapy in Assiut University Hospitals.
Status: Not yet recruiting | Type: Observational
Sponsor: Abdulrahman Mahmoud Bakri Ahmed (Other)
Responsible Party: Sponsor-Investigator, Abdulrahman Mahmoud Bakri Ahmed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Cognition affection WBRT
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Brain Tumors Treated by Whole Brain Radition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Whole Brain Radiotherapy (WBRT) is widely used to manage brain metastases and primary brain tumors, but it frequently leads to cognitive decline, affecting patients' quality of life. Cognitive impairments after WBRT can manifest in various domains, including memory, attention, executive function, and processing speed. These changes are attributed to direct radiation damage to neural tissues, particularly the hippocampus and white matter tracts, as well as secondary effects such as inflammation and vascular injury. Existing literature reports that up to 30% of patients may experience significant cognitive deterioration after WBRT, with the degree of impairment influenced by factors like total radiation dose, fractionation schedule, patient age, and baseline cognitive function. Despite these concerns, there is currently no standardized protocol for assessing cognitive changes in patients undergoing WBRT. Hippocampal avoidance and neuroprotective agents like memantine have shown potential in mitigating cognitive side effects, but their implementation remains inconsistent. Furthermore, routine cognitive assessments are not yet part of standard clinical practice, leading to a reactive rather than proactive approach to managing cognitive decline. This gap in early detection and standardized cognitive monitoring highlights the need for better methods to understand and manage the cognitive consequences of WBRT. Without systematic assessment, cognitive impairments may go unrecognized until they significantly impact daily functioning, emphasizing the importance of addressing this issue to better support patients undergoing whole brain radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (18 years or older)

  * Patients diagnosed with brain metastases or primary brain tumor requiring WBRT.
  * Ability to provide informed consent.

Exclusion Criteria:

* • Pre-existing severe cognitive impairments or psychiatric disorders unrelated to cancer treatment.

  * Significant neurological conditions other than brain metastases.
  * Patients unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with brain tumor primary or secondary receiving WBRT.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of cognitive functions before and after WBRT. | 6 months
  Assessing the cognitive function of the subjects using the Montreal Cognitive Assessment (MoCA) scale
  Purpose: To provide a broader assessment of cognitive abilities, including attention, memory, language, visuospatial skills, and executive function.

SECONDARY OUTCOMES:
Evaluation of differences in cognitive affection between primary and secondary brain lesions | 6 months
  Assessing the cognitive function of the subjects using the Montreal Cognitive Assessment (MoCA) scale Purpose: To provide a broader assessment of cognitive abilities, including attention, memory, language, visuospatial skills, and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelrahman, professor of psychiatry, Study Director — Assiut University; Fadia Attiah, Lecturer of Neuropsychiatry, Study Director — Assiut University